CLINICAL TRIAL: NCT02181868
Title: Comparison of Biodegradable and Titanium Fixation Systems in Mandibular Symphysis or Parasymphysis Solitary Fractures
Status: Approved for marketing | Type: Expanded Access
Sponsor: Louqiang Zhang (Other)
Responsible Party: Sponsor-Investigator, Louqiang Zhang, Department of Stomatology, Tianjin Medical University General Hospital
Organization: Tianjin Medical University General Hospital (Other)
Other Study IDs: CBTF110
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Mandible Fracture; Rigid Internal Fixation; Three-dimensional Finite Element
MeSH Terms: conditions — Mandibular Fractures

INTERVENTIONS:
Other: Biodegradable and titanium fixation used in mandibular fractures.

SUMMARY:
The mandible bears a wide range of mechanical load from the contraction of masticatory muscles, and has a significant function in normal chewing movements. Mandibular fractures are the most common maxillofacial fractures, accounting for 40%-71% of all maxillofacial fracture cases with an average of 62%. The etiology of mandibular fractures mainly includes assaults, road traffic accidents (RTAs), falls, and sports injuries. Although a wide variance exists in the reported percentage of anterior mandible fractures, aggregate analysis approximates these fractures at 17% of all mandibular fractures. The rigid internal fixation (RIF) technique has become a common treatment for mandibular fractures, in which titanium plates are used in the operation. Some patients have to remove the titanium plates in a second operation following bone healing because of sequelae, such as stress shielding. Biodegradable plates and screws have been developed to eliminate the problems associated with titanium fixtures. In this study, we aim to compare the clinical performance between biodegradable and titanium fixation systems after 12 months of follow-up in fixation of mandibular symphysis and parasymphysis solitary fractures. We also investigate the stress distributions of biodegradable and titanium fixation systems at mandibular symphysis solitary fracture on the conditions of intercuspal position, labial teeth occlusion, and premolar and molar occlusion using finite element analysis.

ELIGIBILITY:
Inclusion Criteria:

* Undisplaced and displaced mandibular symphysis and parasymphysis solitary fractures conducted at the department of Oral and Maxillofacial (OMF) Surgery, Tianjin Medical University General Hospital

Exclusion Criteria:

* The exclusion criteria were comminuted fractures
* Diabetes
* Connective tissue diseases
* Patients under the age of 18 and over the age of 60

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Dates: Start 2008-01; Primary Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China